CLINICAL TRIAL: NCT05261204
Title: Transcatheter Aortic Valve Implantation Versus Standard Surgical Aortic Valve Operation for Aortic-Valve Stenosis in Patients at Risk to Severe Valve Obstruction.
Brief Title: Transcatheter Aortic Valve Implantation Versus Standard Surgical Aortic Valve Replacement
Acronym: TAVISAR
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Henri Mondor University Hospital (Other); Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Francesco Nappi, Principal Investigator, Centre Cardiologique du Nord
Other Study IDs: CN-22-25
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Prosthesis Survival; Prosthesis; Cardiac, Heart, Functional Disturbance as Result
MeSH Terms: conditions — Prosthesis Failure | interventions — Transcatheter Aortic Valve Replacement; Sutureless Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transcatheter Aortic Valve Implantation: Patients with aortic-valve stenosis at risk to severe valve obstruction who received TAVI with or without CABG or PCI. Individuals were adequately treated per applicable standards, including for coronary artery disease, LV dysfunction, aortic valve stenosis, and heart failure. Patients enrolled in the studies were NYHA functional class II, III, or outpatient NYHA IV.
  Interventions: Device: Transcatheter Aortic Valve Implantation; Procedure: Bioprothesis; Procedure: Sutureless
- Bioprosthesis: Patients with aortic-valve stenosis at risk to severe valve obstruction who undervent SAVR with the use of bioprosthesis with or without CABG or PCI. Individuals were adequately treated per applicable standards, including for coronary artery disease, LV dysfunction, aortic valve stenosis, and heart failure. Patients enrolled in the studies were NYHA functional class II, III, or outpatient NYHA IV.
  Interventions: Device: Transcatheter Aortic Valve Implantation; Procedure: Bioprothesis; Procedure: Sutureless
- Sutureless: Patients with aortic-valve stenosis at risk to severe valve obstruction who were managed by mean of SAVR with the use of sutureless with or without CABG or PCI. Individuals were adequately treated per applicable standards, including for coronary artery disease, LV dysfunction, aortic valve stenosis, and heart failure. Patients enrolled in the studies were NYHA functional class II, III, or outpatient NYHA IV.
  Interventions: Device: Transcatheter Aortic Valve Implantation; Procedure: Bioprothesis; Procedure: Sutureless

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Patients who are deemed receive TAVI first underwent evaluation of their peripheral arteries before the procedure, in order to separate those eligible for transfemoral placement (TFP) from those who would require transapical placement. Technological advances achieved in the new platforms for the treatment of SHD have allowed the use of reduced size catheters and sheaths in the new armamentarium, favoring the TFP technique. The transcatheter valve (TV) is positioned at the level of the native aortic valve during the final step of valve replacement, when the balloon is inflated within the native valve during a brief period of rapid ventricular pacing. The delivery system i traverses the aorta retrograde over a guidewire from its point of insertion in the femoral artery during the use of TFP. Before balloon inflation, the valve and balloon are collapsed on the catheter and fit within the sheath. After balloon inflation, the calcified native valve is replaced by the expanded TV
  Other Names: Transcatheter Aortic Valve Repacement
Procedure: Bioprothesis — The bioprosthesis is implanted using the SAVR procedure during median sternotomy in extracorporeal circulation. Minimally invasive procedures using a thoracotomy approach and peripheral cannulation have found widespread use.
  Other Names: SAVR
Procedure: Sutureless — The sutureless is implanted using the SAVR procedure during median sternotomy in extracorporeal circulation. Minimally invasive procedures using a thoracotomy approach and peripheral cannulation have found widespread use.
  Other Names: SAVR

SUMMARY:
The mechanical intervention is treating aortic valve stenosis (AVS) which may be performed using the standard open surgical approach for aortic valve replacement (AVR) or transcatheter aortic valve implantation (TAVI). The key question of this study is to establish the difference in all-cause and cause-specific (cardiac vs noncardiac) mortality, all hospitalizations for heart failure within 24 months of follow-up, left ventricular reverse remodeling after adjustment for death, as assessed by means of the left ventricular end-diastolic volume (LVEDV), in patients who received the TAVI vs the standard surgical procedure for AVS.

DETAILED DESCRIPTION:
The target population enrolled in the study includes patients with aortic-valve stenosis at risk to severe valve obstruction who have had TAVI or standard surgical procedure of their aortic valve with or without coronary artery by pass grafting (CABG) or percutaneous coronary intervention (PCI). Individuals were adequately treated per applicable standards, including for coronary artery disease (CAD), left ventricular (LV) dysfunction, AVS, and heart failure (HF). Patients enrolled in the studies were New York Heart Association (NYHA) functional class II, III, or outpatient NYHA IV.

Three groups of patients are included in the study. Patients who were managed with TAVI, patients who received AVR with conventional stented xenograft and recipients of AVR undergoing surgery with the use of sutureless aortic valve.

we calculated that a total of 649 patients per group would be needed for 90% power to show an absolute between-groups difference of 10% in the primary outcome at a two-sided alpha level of 0.02 (corrected alpha level to take into account multiple comparison between 3 groups). In this exhaustive study between 2011 and 2021, we hope to include a total of 6700 patients (2800 in the TAVI group, 3200 patients who received AVR with conventional stented xenograft and 700 patients with the use of sutureless aortic valve).

ELIGIBILITY:
Inclusion Criteria:

* Individuals enrolled in TAVI arm were required to have the predicted risk of operative mortality was ≥ 15% and/or a STS score of ≥ 10. A candidate who did not meet the STS score criteria of ≥ 10 was included in the study if a peer review by at least two surgeon investigators concluded and documented that the patient's predicted risk of operative mortality was ≥ 15%. For all group Senile degenerative aortic valve stenosis with echocardiography derived criteria: mean gradient > 40 mm Hg or jet velocity > 4.0 m/s or an aortic valve area (AVA) of < 0.8 cm2 (or AVA index < 0.5 cm2/m2).

Exclusion Criteria:

* • Patients with evidence of an acute myocardial infarction ≤ 1 month before the intended treatment (defined as Q wave MI, or non-Q wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin level elevation.

  * Blood dyscrasias as defined : leukopenia (WBC < 3000 mm3), acute anemia (Hb < 9 mg%), thrombocytopenia (platelet count < 50,000 cells/mm³), history of bleeding diathesis or coagulopathy.
  * Hemodynamic instability requiring inotropic therapy or mechanical hemodynamic support devices
  * Need for emergency surgery for any reason.
  * Hypertrophic cardiomyopathy with or without obstruction.
  * Severe ventricular dysfunction with LVEF < 20%.
  * Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
  * Active peptic ulcer or upper gastro-intestinal bleeding within the prior 3 months.
  * A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine (Ticlid), or clopidogrel
  * (Plavix), or sensitivity to contrast media, which cannot be adequately pre-medicated.
  * For TAVI arm Native aortic annulus size < 18mm or 25mm as measured by echocardiogram.
  * Subject was offered surgery but refused surgery.
  * Recent (within 6 months) cerebrovascular accident or transient ischemic attack.
  * Renal insufficiency (creatinine > 3.0mg/dL) and/or end stage renal disease requiring chronic
  * dialysis.
  * Life expectancy < 12 months due to non-cardiac co-morbid conditions.
  * For TAVI group significant abdominal or thoracic aorta disease, including aneurysm (defined as maximal luminal diameter 5 cm or greater), marked tortuosity, aortic arch atheroma, narrowing of the abdominal aorta with particular regard for calcification and surface irregularities, or severe "unfolding" and tortuosity of the thoracic aorta. This criteria were applicable for transfemoral patients only.
  * For TAVI group Iliofemoral vessel characteristics that would preclude safe placement of 14F or 18F introducer
  * For TAVI arm sheath such as severe calcification, severe tortuosity or vessels size diameter < 7 mm for 22F
  * Active bacterial endocarditis or other active infections.
  * For TAVI arm bulky calcified aortic valve leaflets in close proximity to coronary ostia.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with aortic valve stenosis with or without CAD who were symptomatic of congestive heart failure and unresponsive to medical therapy and who were eligible for mechanical intervention performed with the use of TAVI procedure or surgical aortic valve replacement. The severity of AVS was assessed by transthoracic echocardiography, performed using the European Society of Echocardiography criteria.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 5 years
  The primary end point of the study is the degree of treatment failure as assessed by death, recurrent aortic valve regurgitation and reoperation
Hospitalizations for Heart Failure (HF) | 5 yeras
  The secondary endpoint of the study is the evaluation of hospedalization rates for heart failure valve due to structural/ non structural valve deterioration, thromboembolism and recurrent endocarditis

SECONDARY OUTCOMES:
Overall Mortality | 5 years
  The secondary endpoint of the study is the evaluation of overall mortality
Cardiac Death | 5 years
  The secondary endpoint of the study is the evaluation of cardiac death
Non Cardiac Death | 5 years
  The secondary endpoint of the study is the evaluation of non cardiac death
Major Adverse Cardiac or Cerebrovascular Events (MACCE) | 5 years
  Composite of major adverse cardiac or cerebrovascular events (rate of death, stroke, subsequent mitral valve surgery, hospitalization for heart failure, or an increase in New York Heart Association class higher than one), serious adverse events, recurrent aortic regurgitation, quality of life, and rehospitalization
Echocardiographic Parameter Changes (LVEF) | 5 years
  Changes from baseline parameters including left ventricular ejection fraction
Echocardiographic Parameter Changes ( AVR recurrence) | 5 years
  Recurrent moderate-to-severe aortic regurgitation after intervention
Echocardiographic Parameter Changes (LVEDD/LVEDV) | 5 years
  Changes from baseline Left Ventricular End Diastolic Diameter or Volume

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, Principal Investigator — Cardiac Surgery Centre Cardiologique du Nord de Saint-Denis, Paris, France
Locations (1):
- Francesco Nappi, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nappi F, Bourgois C, Nenna A, Salsano A, Schoell T, El-Dean Z, Fiore A, Spadaccio C. Study protocol for an internahaational prospective non-randomised trial evaluating the long-term outcomes of transcatheter aortic valve implantation versus surgical aortic valve replacement for aortic-valve stenosis in patients at risk to severe valve obstruction: the TAVISAR trial. BMJ Open. 2025 May 24;15(5):e101417. doi: 10.1136/bmjopen-2025-101417. PMID 40413055